CLINICAL TRIAL: NCT04632914
Title: Effect of Trunk Stabilizing Exercises on Sternal Instability and Separation in Patients With Median Sternotomy After Heart Valve Surgery: A Randomized Clinical Trial
Brief Title: Effect of Trunk Stabilizing Exercises on Patients With Median Sternotomy After Heart Valve Surgery
Acronym: SIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Al Shaymaa Shaaban Abd El Azeim, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/002895
Record Dates: First submitted 2020-10-29; First posted 2020-11-17 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-10

CONDITIONS: Valvular Heart Disease
Keywords: Trunk stabilizing exercises
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Intervention Model Description: trunk stabilizing exercises and cardiac rehabilitation program
Masking Description: no masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- trunk stabilizing exercise (Experimental): trunk stabilizing exercises three times/week for four weeks
  Interventions: Other: trunk stabilizing exercise; Other: cardiac rehabilitation programe
- cardiac rehabilitation programe (Active Comparator): cardiac rehabilitation program three times/week for four weeks
  Interventions: Other: cardiac rehabilitation programe

INTERVENTIONS:
Other: trunk stabilizing exercise — trunk stabilizing exercise is a group of exercise which train the anterior thoracic cage and abdominal muscles in the form of static contraction of these muscles from a different position supine, sitting and standing.
  Arms: trunk stabilizing exercise
Other: cardiac rehabilitation programe — all patients continue this routine physiotherapy program for 40-60min.the patients incorporated into a variety of exercises conducted through arm ergometer,leg ergometer and treadmill.also the patients perform deep breathing exercise and coughing ececise

SUMMARY:
PURPOSE:

The aim of this study is to investigate the effect of trunk stabilizing exercises on sternal instability in patients with median sternotomy after heart valve surgery

DETAILED DESCRIPTION:
Valvular heart disease constitutes a growing healthcare problem with a general prevalence of 2%-5% and a prevalence of 13% after the age of 75 years. Heart valve surgery can be a lifesaving procedure for patients with severe symptomatic heart valve disease. Nevertheless, following the surgery, up to 27% of patients may require readmission within 30 days after discharge. Following heart valve surgery, some patients report anxiety and worries related to readmission and reoperations, postoperative complications, and deconditioning which may prevent or delay return to work and limit activities of daily living Trunk stabilizing exercises train and activate the abdominal and anterior thoracic cage muscles to assist in stabilizing the bisected sternum, thereby decreasing the undue motion in both sagittal and transverse planes during trunk movement. Patients' complaints of pain and discomfort associated with sternal instability post-cardiac surgery may be managed by diminishing the degree of this undue motion between the edges of the divided sternum, and thus provides a conservative treatment for sternal instability forty female patients will be divided into two groups. group A received trunk stabilizing exercise and group B will receive routine cardiac rehabilitation; three times/week for four weeks. the outcome variables were sternal instability and sternal separation and measured before and after completion of treatment

ELIGIBILITY:
Inclusion Criteria:

1. age between 40 and 50 years, female gender
2. hemodynamic stability
3. BMI from 25 to 29.9 kg/m2
4. they will have acute sternal instability.

Exclusion Criteria:

1. previous thoracic surgery
2. elective and urgent coronary artery bypass surgery
3. respiratory insufficiency after surgery manifesting hypoxemia with partial pressure of oxygen in arterial blood <60 mmHg
4. renal insufficiency with serum creatinine ≥1.8 mg/dl after surgery
5. low cardiac output syndrome with ST segment elevation in multiple electrocardiogram leads, cardiac arrhythmias, or hypotension, according to the American College of Cardiology Foundation and American Heart Association
6. other medical conditions such as diabetes, uncontrolled hypertension and obesity
7. Past medical history that include conditions that may have influenced the provision of physiotherapy interventions such as (severe asthma, chronic airflow limitation, bronchiectasis, ankylosing spondylitis or lumbar disc prolapse

Ages: 40 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-11-21 (Estimated); Primary Completion 2020-12-25 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
sternal separation | it will be measured after four weeks
  ultrasound unit will be used to measure the transverse distance between the two edges of stenum

SECONDARY OUTCOMES:
sternal instability | it will be measured after four weeks
  sternal instability scale will be used to assess the integrity of the sternum and transferring the results of the assessment to an acceptable grade

CONTACTS AND LOCATIONS:
Locations (1):
- Al Shaymaa Shaaban Abd El Azeim, Giza, Egypt

REFERENCES:
- [Derived] Essam El-Sayed Felaya ES, Abd Al-Salam EH, Shaaban Abd El-Azeim A. Trunk stabilising exercises promote sternal stability in patients after median sternotomy for heart valve surgery: a randomised trial. J Physiother. 2022 Jul;68(3):197-202. doi: 10.1016/j.jphys.2022.06.002. Epub 2022 Jun 23. PMID 35753968